CLINICAL TRIAL: NCT05863065
Title: Personalized Virtual Reality Naturalistic Scenarios Promoting Engagement and Relaxation in Patients With Cognitive Impairment: a Proof-of-concept Mixed-methods Study
Brief Title: Personalized Virtual Reality Naturalistic Scenarios in Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Fondazione Bruno Kessler (Other); Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento (Other); TrentinoSalute4.0 (Other)
Responsible Party: Principal Investigator, Caterina Novara, Associate Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VR2022
Record Dates: First submitted 2023-04-28; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Impairment; Cognitive Decline; Cognitive Deterioration; Anxiety State
Keywords: virtual reality; personalized virtual scenario; user centered approach; mixed-methods study; user-experience; feasibility study; relaxation; anxiety
MeSH Terms: conditions — Cognitive Dysfunction; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Virtual Reality exposure (Experimental): Participants are exposed to a personalized, relaxing VR scenario administered by the Oculus Quest 2 tool.
  Interventions: Other: Exposure to a Virtual Reality scenarios

INTERVENTIONS:
Other: Exposure to a Virtual Reality scenarios — Exposure to a personalized, relaxing Virtual Reality scenario deployed by a Head-mounted tool (Oculus Quest 2). The administration was deployed in one session.

SUMMARY:
The goal of this feasibility study is to investigate the feasibility of a personalized naturalistic Virtual Reality scenario by assessing motion-sickness effects, engagement, pleasantness, and emotions felt considering a sample of individuals with cognitive impairment resident at the Azienda Pubblica di Servizi alla Persona (APSP) "Margherita Grazioli", a long-term care home in Trento (Italy) in collaboration with the Department of General Psychology - University of Padova (Italy) and the Centre for Health and Wellbeing-Fondazione Bruno Kessler (Italy). The current proof-of-concept and feasibility study is a one-session single-centre trial based on a mixed-methods approach inspired by the Obesity-Related Behavioral Intervention Trials (ORBIT) framework for the design (Phase Ib) of digital interventions and their preliminary testing (Phase IIa).

DETAILED DESCRIPTION:
The impact of customizing VR scenarios is growing, showing different kinds of positive effects, such as an increased sense of presence and engagement in the virtual environment. A relaxing and customizable VR environment could allow the management of any interfering environmental factors that might also be present in the natural context. Additional investigations are still needed to obtain more consistent data on its feasibility and effectiveness.

Considering this evidence, the current proof-of-concept study is based on the following goals:

* evaluate the impact of VR on self-reported and observational levels of motion-sickness, engagement, and pleasantness in older adults living with cognitive impairment and residing in long-term care.
* investigate if personalized, relaxing virtual environments can positively impact feelings and state anxiety.
* investigate the VR apparatus's usability from the health staff's perspective.

ELIGIBILITY:
Inclusion Criteria:

* Italian mother tongue
* Clinical diagnosis of Cognitive Impairment (mild, moderate, or severe).

Exclusion Criteria:

* Palliative care
* Clinical diagnosis of psychosis
* Severe neurological damage
* A clinical diagnosis of epilepsy (or having first-degree relatives diagnosed with epilepsy) - - Cardiac pacemaker or other metal devices
* Infectious or gastrointestinal disorders
* Open wounds at the level of the face
* Motor or visual dysfunctions and neuromuscular pain that prevent the use of Oculus.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Assessing the general and eye-related physical symptoms of exposure to a virtual reality environment. | Through study completion, an average of 6 months
  To assess these symptoms, the Virtual Reality Symptom Questionnaire (VRSQ) was used. The score assigned to each item ranges from 0 to 6, with a maximum total score of 84 (48 for general symptoms and 36 for eye symptoms). Higher scores represent worse symptoms, with 0 corresponding to no adverse effects, and 84 to serious adverse effects.
VR experience tolerability estimated based on the frequency of time spent in the VR context. | Through study completion, an average of 6 months
  The VR experience tolerability was estimated based on the frequency of time spent in the VR context.
Usability of the VR apparatus | Through study completion, an average of 6 months
  The usability has been investigated by a measure developed and described by Appel et al. (2020) composed of both self-reported questions and other queries that the experimenter answered by observing the participant's behavior during the experience and characterized by a series of items based on a 5 points Likert scale (Questions about Level of interest, awareness, engagement, and enjoyment observed: 1="very much", 5="not at all"; min. score=5 and max. score=25; higher scores mean a worse outcome. Questions on other information in relation to the VR experience: 1= "strongly disagree", 5= "strongly agree"; min. score=17 and max. score=85; higher scores mean a better outcome), and six open-ended questions focalized in obtaining additional information, where possible, about: 1) what participants liked best and least; 2) what participants would like to see; 3) if participants would like to repeat the experience; 4) if participants would recommend the experience to a friend.

SECONDARY OUTCOMES:
Change from before and after the one-shot VR session in the relaxation using the modified version of the State-Trait Anxiety Inventory-Y1 (STAI-Y1). | Through study completion, an average of 6 months
  The modified version of the State-Trait Anxiety Inventory-Y1 (STAI-Y1), inspired by Appel et al.16,17, was administered in this study to obtain information on the state-anxiety level experienced before and after the VR session.
  The scale was administered as an interview based on a 5-point Likert scale from 1 (not at all) to 5 (a lot); min. score=15; max. score=75. Higher scores mean a worse outcome.
Change from before and after the one-shot VR session in emotions felt using the Observed Emotion Rating Scale (OERS). | Through study completion, an average of 6 months
  The Observed Emotion Rating Scale (OERS) was adapted from the original version of Lawton et al.41 and used as an observation tool to assess the presence and frequency of negative emotions (fear, anxiety, anger, and sadness) and positive (pleasure) feelings experienced during the session based on a scale from 1 to 5 (1: "undetected emotion"; 2: "emotion observed for less than 16 seconds"; 3: "emotion observed for 16-59 seconds"; 4: "emotion observed for 1-5 minutes"; 5: "emotion observed for more than 5 minutes").
Feedback about the perceived quality rating of the VR set-up deployed from health care staff | Through study completion, an average of 6 months
  To obtain information from health professionals about the perceived quality rating of the VR set-up deployed, the Adapting-Mobile App Rating Scale (A-MARS)-Subjective Quality Scale was filled in by operators who participated during the VR sessions. The administration was performed at the end of the administration of the experimental procedure. (Likert scale from 1 to 5; min.score=4 and max.score=25; higher scores mean a better outcome).
Feedback about usability from health care staff | Through study completion, an average of 6 months
  To obtain information from health professionals about usability of the VR set-up deployed, the System Usability Scale (SUS) was filled in by operators who participated during the VR sessions. The administration was performed after the administration of the experimental procedure. The SUS consists of a 10 item questionnaire on a 5-points Likert scale (1: Strongly agree; 5: Strongly disagree). The score for each question is converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Higher scores mean a better outcome.
Feedback about acceptability from health care staff | Through study completion, an average of 6 months
  To obtain information from health professionals about acceptability, at the end of the experimental phase, a focus group was conducted with the health professionals that assisted users during the VR experience. Issues discussed during the focus group were the strengths and weaknesses associated with using virtual reality, the future perspectives, and the risks associated with using virtual reality with users affected by cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Pardini, PsyD, Principal Investigator — University of Padova; Caterina Novara, PhD, Principal Investigator — University of Padova
Locations (2):
- Italy (2):
  - University of Padova, Padua, PD
  - Azienda Pubblica di Servizi alla Persona (APSP) "Margherita Grazioli", Trento, TN

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pardini S, Gabrielli S, Gios L, Dianti M, Mayora-Ibarra O, Appel L, Olivetto S, Torres A, Rigatti P, Trentini E, Leonardelli L, Bernardi M, Lucianer M, Forti S, Novara C. Customized virtual reality naturalistic scenarios promoting engagement and relaxation in patients with cognitive impairment: a proof-of-concept mixed-methods study. Sci Rep. 2023 Nov 22;13(1):20516. doi: 10.1038/s41598-023-47876-1. PMID 37993549